CLINICAL TRIAL: NCT05649241
Title: Testing the Efficacy, Feasibility and Acceptability of a Pharmacist-Delivered Medication Therapy Management Approach to Smoking Cessation for Rural Smokers in Appalachia
Brief Title: QuitAid Pilot Feasibility Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Melissa Little, PhD, MPH, Associate Professor, Department of Public Health Sciences, University of Virginia
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HSR210262
Record Dates: First submitted 2022-12-04; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Use Cessation Devices; Nicotine; Nicotine Chewing Gum; Medication Therapy Management

STUDY DESIGN:
Intervention Model Description: 2x2x2 factorial design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- QuitAid, 8 weeks, Patch + Gum (Experimental): Participants received QuitAid, a medication therapy management delivered by their pharmacists and 8 weeks of Nicotine Replacement Therapy (NRT) in the form of the NRT Patch and the NRT Gum
  Interventions: Drug: Nicotine patch; Drug: Nicotine gum; Behavioral: Medication Therapy Management
- QuitAid, 4 weeks, Patch + Gum (Experimental): Participants received QuitAid, a medication therapy management delivered by their pharmacists and 4 weeks of Nicotine Replacement Therapy (NRT) in the form of the NRT Patch and the NRT Gum
  Interventions: Drug: Nicotine patch; Drug: Nicotine gum; Behavioral: Medication Therapy Management
- QuitAid, 8 weeks, Patch (Experimental): Participants received QuitAid, a medication therapy management delivered by their pharmacists and 8 weeks of Nicotine Replacement Therapy (NRT) in the form of the NRT Patch
  Interventions: Drug: Nicotine patch; Behavioral: Medication Therapy Management
- QuitAid, 4 weeks, Patch (Experimental): Participants received QuitAid, a medication therapy management delivered by their pharmacists and 4 weeks of Nicotine Replacement Therapy (NRT) in the form of the NRT Patch
  Interventions: Drug: Nicotine patch; Behavioral: Medication Therapy Management
- No QuitAid, 8 weeks, Patch + Gum (Experimental): Participants received 8 weeks of Nicotine Replacement Therapy (NRT) in the form of the NRT Patch and the NRT Gum
  Interventions: Drug: Nicotine patch; Drug: Nicotine gum
- No QuitAid, 4 weeks, Patch + Gum (Experimental): Participants received 4 weeks of Nicotine Replacement Therapy (NRT) in the form of the NRT Patch and the NRT Gum
  Interventions: Drug: Nicotine patch; Drug: Nicotine gum
- No QuitAid, 8 weeks, Patch (Experimental): Participants received 8 weeks of Nicotine Replacement Therapy (NRT) in the form of the NRT Patch
  Interventions: Drug: Nicotine patch
- No QuitAid, 4 weeks, Patch (Experimental): Participants received 4 weeks of Nicotine Replacement Therapy (NRT) in the form of the NRT Patch
  Interventions: Drug: Nicotine patch

INTERVENTIONS:
Drug: Nicotine patch — Nicotine replacement therapy patch
  Other Names: Nicoderm CQ; nicotine transdermal system patch; Habitrol; Nicotrol
Drug: Nicotine gum — Nicotine replacement therapy gum
  Other Names: nicorette; lucy; habitrol; pixotine
  Arms: No QuitAid, 4 weeks, Patch + Gum; No QuitAid, 8 weeks, Patch + Gum; QuitAid, 4 weeks, Patch + Gum; QuitAid, 8 weeks, Patch + Gum
Behavioral: Medication Therapy Management — Medication therapy management delivered by pharmacist - 1 in-person coaching session, and 5 follow-up telephonic coaching sessions.
  Other Names: QuitAid
  Arms: QuitAid, 4 weeks, Patch; QuitAid, 4 weeks, Patch + Gum; QuitAid, 8 weeks, Patch; QuitAid, 8 weeks, Patch + Gum

SUMMARY:
Adult smokers were recruited through an independent pharmacy in rural Appalachia and were randomized to 1 of 8 treatments, including medication and/or therapy from the pharmacist, to help quit smoking.

DETAILED DESCRIPTION:
24 adult smokers were recruited through an independent pharmacy in rural Appalachia were randomized to 1 of 8 treatments: (1) pharmacist delivered QuitAid intervention (Yes vs. No), (2) Combination NRT Gum + NRT Patch (vs. NRT patch), and/or (3) 8 weeks of NRT (vs. standard 4 weeks). All participants received 4 weeks of NRT patch in addition to the components to which they were assigned. Participants completed baseline and 3-month follow-up assessments. The primary outcomes were feasibility of recruitment and randomization, retention, treatment adherence and fidelity.

ELIGIBILITY:
Inclusion Criteria:

* smokers must have smoked at least 5 cigarettes per day for the past 6 months
* be willing to set a quit date in the next 30 days
* own a cell phone
* be over 18 years of age
* not be pregnant or planning to become pregnant in the next 6 months
* not have any medical contraindications to using NRT

Exclusion Criteria:

* Those who are pregnant or plan to be
* Those under 18 years of age
* Those with a medical contradiction
* Those who do not own a cell phone
* Those who have not smoked 5 cigarettes per day for the last 6 months
* Those who are unwilling to set a quit date within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment | 3 months
  Feasibility of recruitment was measured by (a) the proportion of smokers recruited from each source (e.g., ask-advise-connect, posters, prescription bag advertisements) and (b) the number recruited per month.
Feasibility of randomization | 3 months
  Feasibility of randomization was determined by the number of smokers that were approached and screened in order to randomize 24 smokers (e.g., ineligible smokers, smokers that do not consent).
Retention | 3 months
  Retention was assessed by the proportion of smokers who completed the 3-month follow-up.

SECONDARY OUTCOMES:
Tobacco Use | 3 months
  Biochemically verified self-reported point prevalence tobacco abstinence at the 3-month follow-up was collected

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Little, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Little MA, Reid T, Moncrief M, Cohn W, Wiseman KP, Wood CH, You W, Anderson RT, Krukowski RA. Testing the feasibility of the QuitAid smoking cessation intervention in a randomized factorial design in an independent, rural community pharmacy. Pilot Feasibility Stud. 2024 Feb 26;10(1):41. doi: 10.1186/s40814-024-01465-9. PMID 38409089